CLINICAL TRIAL: NCT02234193
Title: A Pilot Clinical Trial to Reduce Side-effects of Autologous Skin Tissue Harvesting
Brief Title: Reducing Side-effects of Autologous Skin Tissue Harvesting
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Richard Rox Anderson, MD, Professor of Dermatology, Director of the Wellman Center for Photomedicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014P000120
Record Dates: First submitted 2014-08-27; First posted 2014-09-09 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Scar
Keywords: wound healing
MeSH Terms: conditions — Cicatrix | interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Micro biopsies 2mm x control (Active Comparator): 2 mm diameter micro biopsies will be performed on all subjects.
  Interventions: Device: Micro biopsy; Procedure: Lidocaine with epinephrine
- Micro biopsies 1mm x control (Active Comparator): 1 mm diameter micro biopsies will be performed on all subjects.
  Interventions: Device: Micro biopsy; Procedure: Lidocaine with epinephrine
- Micro biopsies 0.8 mm x control (Active Comparator): 0.8 mm diameter micro biopsies will be performed on all subjects.
  Interventions: Device: Micro biopsy; Procedure: Lidocaine with epinephrine
- Micro biopsies 0.6 mm x control (Active Comparator): 0.6 mm diameter micro biopsies will be performed on all subjects.
  Interventions: Device: Micro biopsy; Procedure: Lidocaine with epinephrine
- Micro biopsies 0.5 mm x control (Active Comparator): 0.5 mm diameter micro biopsies will be performed on all subjects.
  Interventions: Device: Micro biopsy; Procedure: Lidocaine with epinephrine
- Micro biopsies 0.40 mm x control (Active Comparator): 0.4 mm diameter micro biopsies will be performed on all subjects.
  Interventions: Device: Micro biopsy; Procedure: Lidocaine with epinephrine
- Micro biopsies 0.20 mm x control (Active Comparator): 0.2 mm diameter micro biopsies will be performed on all subjects.
  Interventions: Device: Micro biopsy; Procedure: Lidocaine with epinephrine

INTERVENTIONS:
Device: Micro biopsy — This is a prospective, self-controlled study of the healing response after collecting micro skin biopsies of different sizes (from 200 µm to 2 mm in diameter) from up to seven 1.5 x 1.5 cm biopsy sites in pre-abdominoplasty skin areas that are scheduled for surgical removal. The collection procedure will be performed using similar techniques as standard skin biopsies: the skin area involved will be cleaned with alcohol pads, and 1% buffered lidocaine with epinephrine anesthesia will be administered locally, then micro biopsies of skin will be removed by biopsy punch/harvesting needle. No more than 10% of the skin area within each biopsy site will be collected. Tattoo ink as described will be applied to 4 micro-biopsies at the corners of each biopsy test site
Procedure: Lidocaine with epinephrine — The skin area involved will be cleaned with alcohol pads, and 1% buffered lidocaine with epinephrine anesthesia will be administered locally, prior to the surgical procedure
  Other Names: Lidocaine

SUMMARY:
The investigators are doing this research study to learn about how the skin heals after many microscopic skin biopsies are collected.

Skin-grafting is a life-saving procedure for people with large area skin wounds caused by burns or trauma. Conventional autologous (self) skin grafting techniques require the creation of large donor site wounds, causing numerous complications including pain, infection, blistering, discoloration, and scarring. Based on previous research, many of these adverse effects can be improved, or even eliminated, by harvesting skin tissue in very small biopsies. These "micro-biopsies" are less than the size of a sewing pin. Then, they are put back together into a skin graft.

This concept is based on clinical observations from fractional photothermolysis laser therapy, an FDA approved laser that has been previously developed by the investigators research group for the treatment of scars and ageing skin. With this laser technique, thousands to millions of small burns are produced by laser on a patient's skin, and the skin responds by healing the damaged areas to create new healthy skin within days and without scarring.

Although the results of laser treatment are well-known, it is not known what happens when we harvest the skin using needles instead of using the laser to cut the skin. The investigators also would like to understand how the body heals the skin. Understanding how this works helps in understanding wound healing, and may lead to future treatments for healing large wounds, disfiguring burn scars, and preventing scar formation.

A tummy tuck (abdominoplasty surgery) is done to remove excessive skin of the belly. This is an elective surgery, in other words, it is optional and usually done for cosmetics reasons (to improve the appearance).

The skin of the belly that is removed during an abdominoplasty surgery (tummy tuck) is discarded. The skin of the area removed is called "pre-abdominoplasty skin". The investigators would like to study the effects of the micro-biopsies on pre-abdominoplasty skin to exam how the skin heals over time and to study the skin that will be removed during the abdominoplasty surgery.

This is a pilot study. Pilot studies are done on a small group of subjects to learn if a larger study would be useful.

The investigators are asking subjects to take part in this study who are healthy with an abdominoplasty surgery (tummy tuck) scheduled at Massachusetts General Hospital (MGH) by a plastic surgeon .

The investigators will enroll about 28 subjects in this research study, all at MGH.

The Department of Defense is paying for this study to be done.

DETAILED DESCRIPTION:
It will take you about 8 weeks to complete this research study. During this time, the investigators will ask you to make up to 7 study visits to MGH.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults (>18 years old) scheduled to undergo elective abdominoplasty surgery at MGH, male or female.
2. Willingness to participate in the study
3. Willingness to undergo biopsies of full-thickness skin tissue from the pre-abdominoplasty skin, and have the biopsy sites marked by tattoos.
4. Informed consent agreement signed by the subject
5. Willingness to follow the treatment and follow-up schedules, and post treatment care requirements
6. Willingness to not use topical or systemic (oral) anti-scarring or anti-inflammatory* medications during the study period.

Exclusion Criteria:

1. Subjects who are immunocompromised or immunosuppressed*
2. Subject is unable to comply with treatment, home care or follow-up visits
3. Subject has an infection or other dermatologic condition in the area to be treated
4. Subjects with a personal or family history of keloid formation.
5. Subjects with pre-existing scars, tattoos, birthmarks, or other physical features in the area to be treated, such that the experimental outcome may be confounded.
6. Subjects with a history of coagulopathy, or are taking anticoagulants
7. Subjects taking daily oral aspirin.
8. Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
9. Subjects with any contraindications for elective abdominoplasty, as determined by their treating plastic surgeon and/or pre-op anesthesiologist.
10. Subjects with current drug or alcohol addiction.
11. Subjects who are pregnant and/or breastfeeding
12. Subjects with tape adhesive allergies
13. Subjects with known allergies to injectable lidocaine or other topical anesthetics
14. Subjects with uncontrolled or unstable chronic disease such as diabetes, hepatitis, hypertension, etc.
15. Subjects taking oral corticosteroids or topical steroids on the study area.
16. Subjects using prescription or over-the-counter medication or cosmetics containing: retinoids, glycolic acid, salicylic acid or any other remedies that might affect the healing process. (Non-medicated moisturizers are ok).
17. Subjects enrolled in other clinical studies taking any unknown or not-FDA approved medications.
18. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Notes:

*About Anti-Inflammatory Medication and Immune Status The inflammatory response associated with tissue wounding is known to have substantial effects on the process of scarring, therefore all subjects who are immunocompromised, or undergoing anti-inflammatory/immunosuppressive therapies will be excluded from the study. All new medication should be reported to study doctor before each visit.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of Efficacy - Change from baseline scarring at 8 weeks | 24 h, 1 week, 2 weeks, 4 weeks and 8 weeks post treatment
  The extent of scarring caused by the harvesting of micro-skin columns will be assessed by investigators and patients using the Patient and Observer Scar Assessment Scale (POSAS) at all of the follow-up time points.
  Patient and Observer Scar Assessment Scale (POSAS)

SECONDARY OUTCOMES:
Assessing Subject Side-effects - Change from baseline side-effects at 8 weeks | day 0, 24 h, 1 week, 2 weeks, 4 weeks and 8 weeks after the procedure
  A Major side effect is defined as an intolerable side effect that would warrant the cessation of treatment because of a risk to the subject's health or because the subject could not tolerate the treatment due to a subjective personal measure (e.g. severe pain). A Minor side effect is a side effect that while uncomfortable would not threaten the subject's health or cause the cessation of treatment due to lack of comfort.
  Major side effects include: severe pain (Pain ≥ 8/10 on VAS scale), severe blistering (with potential for secondary infection) and ulceration with scarring. Subjects will be asked for each site to fill in the following sentence: "The side effects I experienced with micro biopsies were: "0: Did not have this side effect / 1: Mild / 2: Moderate / 3: Severe Swelling, Redness, Scabs, Pus or pus blisters, Scaling, Itchy skin, Erosion, Tanning, Lightening of the skin, Minor blistering, Wheals, Bleeding, Folliculitis, Oozing, Numbness
Pain assessment - Visual Analog Scale (VAS) - Change from baseline pain at 8 weeks | DAY 0, 24h, 1, 2, 4 & 8 weeks
  The VAS will be completed by study subject at baseline and at each follow-up visit for each test site.
  Pain is any of the following: sensation of tingling, stinging, prickling, or burning feeling, heat under the skin, tenderness, mild, moderate or severe pain).
  Specific VAS form is attached
  Subjects will be asked to circle the number below that most closely corresponds to pain associated with each treatment site.
  0 1 2 3 4 5 6 7 8 9 10 (NO PAIN WORST PAIN)

OTHER OUTCOMES:
Histopathology examination | 8 weeks
  After the subject's elective abdominoplasty procedure, the excised skin will be collected. Samples will be taken from the excised skin in areas where micro skin biopsies were harvested at time 0 (visit 2). Since all tissue samples are collected from skin that has already been excised during abdominoplasty surgery, the collection of samples for histopathology poses no additional risk for the subjects.
Subject Satisfaction Survey - Change from baseline side-effects at 8 weeks | Day 0, 24h, 1, 2, 4 & 8 Weeks
  In this survey, subjects are given a list of the side effects of the micro-biopsies before treatment (Visits1-7) and are asked to rate each question on a scale of 1 to 5. After treatment, they are given this specific survey (but specific to each treatment site) after each month of treatment as a repeated measure of side effects, before and after each procedure. They will be asked the question based on the treatment site name, if they consider the treatment cosmetically acceptable. For example:
  Answer the questions bellow with a number:
  5 Agree Strongly 4 Agree 3 Neutral 2 Disagree 1 Disagree Strongly The treatment performed on the SITE 1 (same for other sites SITES) SITE 1 treatment is safe SITE 1 treatment is cosmetically sound (Do you think it looks ok?). The side effects of SITE 1 treatment are tolerable.

CONTACTS AND LOCATIONS:
Locations (1):
- Wellman Center for Photomedicine, Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Rasmussen CA, Tam J, Steiglitz BM, Bauer RL, Peters NR, Wang Y, Anderson RR, Allen-Hoffmann BL. Chimeric autologous/allogeneic constructs for skin regeneration. Mil Med. 2014 Aug;179(8 Suppl):71-8. doi: 10.7205/MILMED-D-13-00480. PMID 25102552
- [Derived] Champlain AH, DiGiorgio CM, Zurakowski D, Sakamoto FH, Anderson RR. Wound Healing After Fractional Skin Harvesting. Dermatol Surg. 2022 Oct 1;48(10):1083-1088. doi: 10.1097/DSS.0000000000003552. Epub 2022 Aug 23. PMID 36036977